CLINICAL TRIAL: NCT00251459
Title: A Phase IIIb, Single-Masked, Multicenter, Randomized Study to Evaluate the Safety and Tolerability of Ranibizumab in Naive and Previously Treated Subjects With Choroidal Neovascularization (CNV) Secondary to Age-Related Macular Degeneration (AMD)
Brief Title: A Study to Evaluate Ranibizumab in Subjects With Choroidal Neovascularization (CNV) Secondary to Age-Related Macular Degeneration (AMD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Purpose: Treatment
Other Study IDs: FVF3689g; NCT00299078 (obsolete NCT alias)
Record Dates: First submitted 2005-11-08; First posted 2005-11-10 (Estimated); Last update posted 2014-03-10 (Estimated); Status verified 2014-03

CONDITIONS: Choroidal Neovascularization; Age-related Macular Degeneration
Keywords: SAILOR; CNV; AMD; CNV secondary to AMD
MeSH Terms: conditions — Choroidal Neovascularization; Macular Degeneration | interventions — Ranibizumab

INTERVENTIONS:
Drug: rhuFab V2 (ranibizumab)

SUMMARY:
This is a Phase IIIb, single-masked, 1-year multicenter study of the safety and tolerability of intravitreally administered ranibizumab in subjects with active subfoveal CNV secondary to AMD.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent Form
* Age ≥ 50 years
* Subfoveal CNV secondary to AMD, with evidence of recent disease progression, as defined by any of the following (lesion is eligible if it meets any one of the following criteria): ≥ 5 letters (or ≥ 1 Snellen line) of BCVA lost within 6 months preceding Day 0\; ≥ 10% increase in lesion area, as determined by comparing a FA performed within 1 month preceding Day 0 to a FA performed within 6 months preceding Day 0; Subretinal hemorrhage associated with CNV within 1 month preceding Day 0; Classic CNV comprising > 50% of CNV lesion area
* BCVA, using ETDRS charts for Cohort 1 and Snellen charts for Cohort 2, of 20/40 to 20/320 (Snellen equivalent) in the study eye

Exclusion Criteria:

* Treatment with verteporfin PDT, pegaptanib sodium, or other AMD therapy in the study eye < 30 days preceding Day 0
* History of submacular surgery or other surgical intervention for AMD in the study eye
* Previous participation in any studies of investigational drugs within 30 days preceding Day 0 (excluding vitamins and minerals)
* Prior participation in a Genentech ranibizumab clinical trial
* Treatment with intravitreally administered (in either eye) Avastin(R) (bevacizumab) within 30 days preceding Day 0
* Concurrent use of systemic anti-VEGF agents
* Fibrosis or atrophy involving the center of the fovea in the study eye, in the absence of a new lesion
* CNV in either eye due to other causes, such as ocular histoplasmosis, trauma, or pathologic myopia
* Retinal pigment epithelial tear involving the macula in the study eye
* Any concurrent intraocular condition in the study eye (e.g., cataract or diabetic retinopathy) that, in the opinion of the investigator, could either require medical or surgical intervention during the 12-month study period to prevent or treat visual loss that might result from that condition, or, if allowed to progress untreated, could likely contribute to loss of at least 2 Snellen equivalent lines of BCVA over the 12-month study period
* Active intraocular inflammation (grade trace or above) in the study eye
* Current vitreous hemorrhage in the study eye
* History of rhegmatogenous retinal detachment or macular hole (Stage 3 or 4) in the study eye
* History of idiopathic or autoimmune-associated uveitis in either eye
* Active infectious conjunctivitis, keratitis, scleritis, or endophthalmitis in either eye
* Aphakia or pseudophakia with absence of the posterior capsule (unless it occurred as a result of a yttrium aluminum garnet [YAG] posterior capsulotomy)
* Spherical equivalent of the refractive error in the study eye demonstrating more than -8 diopters of myopia
* Intraocular surgery (including cataract surgery) in the study eye within 2 months preceding Day 0
* Uncontrolled glaucoma in the study eye (defined as intraocular pressure ≥ 25 mmHg despite treatment with antiglaucoma medication)
* Concurrent use of more than one therapy for glaucoma
* History of glaucoma filtering surgery in the study eye
* History of corneal transplant in the study eye
* Premenopausal women not using adequate contraception
* Pregnancy or lactation
* History of other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use an investigational drug or that might affect interpretation of the results of the study or render the subject at high risk for treatment complications
* Current treatment for a significant active systemic infection
* Evidence of significant uncontrolled concomitant diseases such as cardiovascular disease, nervous system, pulmonary, renal, hepatic, endocrine, or gastrointestinal disorders
* History of recurrent significant infections or bacterial infections
* Inability to comply with study or follow-up procedures

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5000
Dates: Start 2005-11; Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Cohort 1: The primary safety outcome measure is the incidence of SAEs (ocular and non ocular) evaluated through Month 12.
Cohort 2: The primary safety outcome measure is the incidence of SAEs (ocular and non-ocular) and AEs (ocular and non-ocular) evaluated through Month 12.

SECONDARY OUTCOMES:
Incidence of AEs (ocular and non-ocular) evaluated through Month 12
Proportion of subjects who lose at least 15 letters in BCVA at Month 12 compared with baseline
Mean time to retreatment following the initial three monthly loading doses
Mean total number of injections through Month 12.

CONTACTS AND LOCATIONS:
Overall Officials: Tsontcho Ianchulev, M.D., Study Director — Genentech, Inc.

REFERENCES:
- [Result] Boyer DS, Heier JS, Brown DM, Francom SF, Ianchulev T, Rubio RG. A Phase IIIb study to evaluate the safety of ranibizumab in subjects with neovascular age-related macular degeneration. Ophthalmology. 2009 Sep;116(9):1731-9. doi: 10.1016/j.ophtha.2009.05.024. Epub 2009 Jul 29. PMID 19643495